CLINICAL TRIAL: NCT00825370
Title: Protocolized vs Discretionary Use of Opioids in Acute Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Andrew Chang, MD, MD, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MMC 0808278
Record Dates: First submitted 2009-01-19; First posted 2009-01-21 (Estimated); Results first posted 2018-04-19 (Actual); Last update posted 2018-06-12 (Actual); Status verified 2018-05

CONDITIONS: Pain
Keywords: Hydromorphone; acute pain; Protocolized; Efficacy; Safety
MeSH Terms: conditions — Pain; Acute Pain | interventions — Hydromorphone; Analgesics, Opioid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Protocolized (Experimental): 1 mg IV hydromorphone followed by an optional 1 mg IV hydromorphone 15 minutes later if the patient answers yes to the question, "Do you want more pain medication?"
  Interventions: Drug: Hydromorphone
- Discretionary Care (Active Comparator): Patients receive an IV opioid the type and dose of which is determined by the treating physician
  Interventions: Drug: IV opioid

INTERVENTIONS:
Drug: Hydromorphone — 1 mg IV hydromorphone followed by an optional 1mg IV hydromorphone 15 minutes later
  Other Names: Dilaudid
  Arms: Protocolized
Drug: IV opioid — Any IV opioid in the dose chosen by the treating physician. May include hydromorphone as well.
  Other Names: Discretionary care
  Arms: Discretionary Care

SUMMARY:
We are testing whether patients who received protocolized pain management (1 mg of IV hydromorphone followed by an additional 1 mg Intravenous (IV) hydromorphone 15 minutes later if the patients wants more) will have better pain relief and no more adverse events than patients receiving discretionary care, in which the patients receives whatever IV opioid the treating physician wants to give, in whatever dose.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21 to 64 years.
2. Pain with onset within 7 days.
3. Emergency Department attending physician's judgment that patient's pain warrants use of intravenous opioids.
4. Normal mental status.

Exclusion Criteria:

1. Prior use of methadone.
2. Use of other opioids, tramadol, or heroin in the past seven days.
3. Prior adverse reaction to morphine, hydromorphone, or other opioids.
4. Chronic pain syndrome.
5. Alcohol intoxication.
6. Systolic Blood Pressure < 90 mm Hg.
7. Use of monoamine oxidase (MAO) inhibitors in past 30 days.
8. Weight less than 100 pounds.
9. Baseline room air oxygen saturation less than 95%.
10. C02 measurement greater than 46: In accordance with a number of similar studies that we have performed, four subsets of patients will have their CO2 measured using a handheld capnometer prior to enrollment in the study. If the CO2 measurement is greater than 46, then the patient will be excluded from the study. The 4 subsets are as follows:

    1. All patients who have a history of chronic obstructive pulmonary disease (COPD)
    2. All patients who have a history of sleep apnea
    3. All patients who report a history of asthma together with greater than a 20 pack-year smoking history
    4. All patients reporting less than a 20 pack-year smoking history who are having an asthma exacerbation

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 350 (Actual)
Dates: Start 2008-10 (Actual); Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew K Chang, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center Emergency Department, The Bronx, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Protocolized | Discretionary Care
Started | 175 | 175
Completed | 175 | 175
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The discrepancy between the number of patients who completed the study and the number of patients included in analysis is due to missing data (6 Protocolized and 4 Discretionary) and participants enrolled more than once (2 Protocolized). These patients completed the study but had duplicate or missing data that could not be included in analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Protocolized | Discretionary Care | Total
Number analyzed (Participants) | 167 | 171 | 338
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (11) | 42 (13) | 42 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107 | 98 | 205
  Male | 60 | 73 | 133
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Hispanic | 110 | 114 | 224
  Race/Ethnicity: Black | 47 | 43 | 90
  Race/Ethnicity: White | 7 | 9 | 16
  Race/Ethnicity: Other | 3 | 5 | 8
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 167 | 171 | 338
Weight [Mean (Standard Deviation); unit: pounds] | 185 (52) | 173 (44) | 179 (48)
Location of pain [Count of Participants; unit: Participants]
  Abdomen | 113 | 95 | 208
  Other | 54 | 76 | 130
Pain Intensity [Count of Participants; unit: Participants] — Pain intensity is measured on a numerical rating score (NRS) scale of 0 ("no pain") to 10 ("worst pain imaginable"). This pain intensity measure is the pain intensity of the patient before treatment in the Emergency Department.
  Participants
    3-7 | 22 | 24 | 46
    8 | 22 | 32 | 54
    9 | 25 | 24 | 49
    10 | 98 | 91 | 189
Nausea [Count of Participants; unit: Participants] | 62 | 44 | 106
Vomiting [Count of Participants; unit: Participants] | 46 | 46 | 92

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Successful Treatment
Description: Successful treatment was defined as either declining additional pain medication when asked at 15 minutes or accepting additional pain medication at 15 minutes but then declining additional pain medication at 60 minutes
Time Frame: 60 minutes
Population: The discrepancy between the number of patients enrolled and randomized and the number of patients included in analysis is due to missing data (6 from Protocolized and 4 from Discretionary Care) and participants enrolled more than once (2 from Protocolized).
Measure: Number; unit: Percentage of Participants
Arm/Group | Protocolized | Discretionary Care
Number analyzed (Participants) | 167 | 171
Percentage of Participants | 86.8 | 76.6

2. Secondary Outcome: Percentage of Patients Who Did Not Want Additional Pain Medication at 15 Minutes
Description: As defined by the percentage of patients who answer "no" to the question, "Do you want more pain medication?" at 15 minutes
Time Frame: 15 min
Measure: Number; unit: Percentage of Participants
Arm/Group | Protocolized | Discretionary Care
Number analyzed (Participants) | 167 | 171
Percentage of Participants | 73.7 | 66.7

3. Secondary Outcome: Percentage of Patients Who Did Not Want Additional Pain Medication at 60 Minutes
Description: Patients who did not want pain medication determined by those who answered "no" to the question "do you want more pain medication?" at 60 minutes after treatment.
Time Frame: 60 minutes
Measure: Number; unit: percentage of participants
Arm/Group | Protocolized | Discretionary Care
Number analyzed (Participants) | 167 | 171
percentage of participants | 72.5 | 63.7

4. Secondary Outcome: Changes in Pain Intensity From Baseline to Other Pain Assessment Times (15 and 60 Minutes).
Description: Mean change in pain intensity between baseline and 15 minutes and between baseline and 60 minutes post treatment. Pain intensity is measured on a numerical rating scale (NRS) from 0 ("no pain") to 10 ("worst pain imaginable"). The averages were calculated by finding the mean of change in pain intensity for each patient.
Time Frame: Up to 60 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Protocolized | Discretionary Care
Number analyzed (Participants) | 167 | 171
units on a scale
  15 minutes | 4.90 (3.1) | 4.55 (3.0)
  60 minutes | 5.32 (3.1) | 4.66 (3.1)

ADVERSE EVENTS:
Time Frame: 60 minutes
Arm/Group | Protocolized | Discretionary Care
All-Cause Mortality (participants affected / at risk) | 0/167 | 0/171
Serious Adverse Events (participants affected / at risk) | 0/167 | 0/171
Other Adverse Events (participants affected / at risk) | 22/167 | 30/171
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Protocolized (N=167) | Discretionary Care (N=171)
Administration of Naloxone (Endocrine disorders) | 0 | 0
Oxygen saturation <95% (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Systolic blood pressure <90 mmHg (Vascular disorders) | 3 | 2
Respiratory rate <12 breaths/min (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 4
Nausea (Gastrointestinal disorders) | 5/82 | 15/102 — excludes patients nauseated before intervention
Vomiting (Gastrointestinal disorders) | 8/120 | 5/125 — excludes patients vomiting before the intervention

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes